CLINICAL TRIAL: NCT02197078
Title: Active Surveillance Research Program for the Assessment of the Safety and the Effectiveness of Linagliptin
Status: Completed | Type: Observational
Sponsor: Boehringer Ingelheim (Industry)
Collaborators: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Other Study IDs: 1218.163
Record Dates: First submitted 2014-07-21; First posted 2014-07-22 (Estimated); Results first posted 2020-04-02 (Actual); Last update posted 2020-04-02 (Actual); Status verified 2020-03

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

GROUPS / COHORTS (4):
- Glitazones
- Linagliptin
- Sulfonylurea
- Within-class comparators

SUMMARY:
This protocol is for a series of comparative effectiveness and safety analyses within periodically updated cohorts of patients initiating linagliptin, other DPP-4 inhibitors, and other oral hypoglycemic medications, followed longitudinally for the occurrence of a variety of health outcomes. The primary analysis will be conducted among patients without prior within-class medication use.

ELIGIBILITY:
Inclusion criteria:

* A dispensing of an oral hypoglycemic medication
* A diagnosis of type 2 diabetes mellitus (T2DM)

Exclusion criteria:

* less than 18 years old
* missing or ambiguous age or sex information
* at least one diagnosis of type 1 diabetes mellitus
* less than 6 months enrolment in the database preceding the date of the first dispensing
* secondary diabetes
* history of cancer
* end-stage renal disease (ESRD)
* HIV
* organ transplant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: T2DM patients aged 18 or older, initiating antidiabetic treatment after at least 6 months of continuous enrollment
Sampling Method: Non-Probability Sample
Enrollment: 189426 (Actual)
Dates: Start 2014-07-30 (Actual); Primary Completion 2019-02-26 (Actual); Study Completion 2019-02-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: From Clinformatics and MarketScan source data, patients with a recorded diagnosis of type 2 diabetes mellitus (T2DM) who initiated linagliptin, sitagliptin, saxagliptin, alogliptin, pioglitazone, or 2nd generation sulfonylureas were identified between May 2011 and December 2016.
Pre-assignment Details: Only participants with no use of a medication in the same class or comparator class during the 6 months prior to index date, who were at least 18 years of age and enrolled for a minimum of 6 months in the data source before treatment initiation were included.
Groups:
- Other DPP-4I - Clinformatics; Linagliptin 1 - Clinformatics: 1:1 propensity score matched cohort of initiators of other Dipeptidyl peptidase-4 (DPP-4) and initiators of linagliptin, within Clinformatics database
- Pioglitazone - Clinformatics; Linagliptin 2 - Clinformatics: 1:1 propensity score matched cohort of initiators of pioglitazone and initiators of linagliptin, within Clinformatics database
- 2nd Gen SUs - Clinformatics; Linagliptin 3 - Clinformatics: 1:1 propensity score matched cohort of initiators of second generation sulfonylureas (2nd gen SUs) and initiators of linagliptin, within Clinformatics database
- Other DPP-4I - MarketScan; Linagliptin 1 - MarketScan: 1:1 propensity score matched cohort of initiators of other Dipeptidyl peptidase-4 (DPP-4) and initiators of linagliptin, within MarketScan database
- Pioglitazone - MarketScan; Linagliptin 2 - MarketScan: 1:1 propensity score matched cohort of initiators of pioglitazone and initiators of linagliptin, within MarketScan database
- 2nd Gen SUs - MarketScan; Linagliptin 3 - MarketScan: 1:1 propensity score matched cohort of initiators of second generation of sulfonylureas (2nd gen SUs) and initiators of linagliptin, within MarketScan database
Period: Overall Study
Arm/Group | Other DPP-4I - Clinformatics | Linagliptin 1 - Clinformatics | Pioglitazone - Clinformatics | Linagliptin 2 - Clinformatics | 2nd Gen SUs - Clinformatics | Linagliptin 3 - Clinformatics | Other DPP-4I - MarketScan | Linagliptin 1 - MarketScan | Pioglitazone - MarketScan | Linagliptin 2 - MarketScan | 2nd Gen SUs - MarketScan | Linagliptin 3 - MarketScan
Started | 14688 | 14688 | 10614 | 10614 | 9538 | 9538 | 25135 | 25135 | 18996 | 18996 | 15742 | 15742
Completed | 14688 | 14688 | 10614 | 10614 | 9538 | 9538 | 25135 | 25135 | 18996 | 18996 | 15742 | 15742
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Participants, who initiated linagliptin, other DPP-4, pioglitazone, or second generation sulfonylureas, were identified from Clinformatics and MarketScan between May 2011 and December 2016.Within each database, a 1:1 propensity score matching was performed between initiators of linagliptin and intiators of each comparator group.
Groups:
- Total: Total of all reporting groups
Arm/Group | Other DPP-4I - Clinformatics | Linagliptin 1 - Clinformatics | Pioglitazone - Clinformatics | Linagliptin 2 - Clinformatics | 2nd Gen SUs - Clinformatics | Linagliptin 3 - Clinformatics | Other DPP-4I - MarketScan | Linagliptin 1 - MarketScan | Pioglitazone - MarketScan | Linagliptin 2 - MarketScan | 2nd Gen SUs - MarketScan | Linagliptin 3 - MarketScan | Total
Number analyzed (Participants) | 14688 | 14688 | 10614 | 10614 | 9538 | 9538 | 25135 | 25135 | 18996 | 18996 | 15742 | 15742 | 189426
Age, Continuous [Mean (Standard Deviation); unit: Years] | 56.31 (12.45) | 56.30 (12.35) | 56.53 (12.48) | 56.77 (12.54) | 55.03 (12.18) | 55.00 (12.21) | 55.25 (11.26) | 55.27 (11.36) | 54.71 (11.22) | 54.73 (11.28) | 54.41 (11.28) | 54.40 (11.31) | 55.39 (11.83)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6118 | 6098 | 4266 | 4337 | 3985 | 3968 | 10377 | 10309 | 7805 | 7850 | 6527 | 6582 | 78222
  Male | 8570 | 8590 | 6348 | 6277 | 5553 | 5570 | 14758 | 14826 | 11191 | 11146 | 9215 | 9160 | 111204
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Major Adverse Cardiovascular Event
Description: Number of participants with major adverse cardiovascular event is presented by the number of patients reported a composite of:
  * Coronary revascularization (elective and non-elective procedure)
  * Acute coronary syndrome (ACS), including acute myocardial infarction (MI)
  * Stroke (Ischemic and hemorrhagic stroke)
Time Frame: Up to 5 years and 7 months
Population: 1:1 propensity score matched cohorts of linagliptin initiators and comparator groups initiators, identified from Clinformatics and MarketScan database between May 2011 and December 2016
Measure: Number; unit: Participants
Arm/Group | Other DPP-4I - Clinformatics | Linagliptin 1 - Clinformatics | Pioglitazone - Clinformatics | Linagliptin 2 - Clinformatics | 2nd Gen SUs - Clinformatics | Linagliptin 3 - Clinformatics | Other DPP-4I - MarketScan | Linagliptin 1 - MarketScan | Pioglitazone - MarketScan | Linagliptin 2 - MarketScan | 2nd Gen SUs - MarketScan | Linagliptin 3 - MarketScan
Number analyzed (Participants) | 14688 | 14688 | 10614 | 10614 | 9538 | 9538 | 25135 | 25135 | 18996 | 18996 | 15742 | 15742
Participants | 165 | 151 | 120 | 102 | 127 | 82 | 403 | 369 | 262 | 270 | 259 | 194
Statistical Analysis 1: Comparison: Other DPP-4I - Clinformatics vs Linagliptin 1 - Clinformatics; Test type: Other; Hazard Ratio (HR) = 0.82, 95% CI 2-sided [0.66 to 1.03]
Statistical Analysis 2: Comparison: Pioglitazone - Clinformatics vs Linagliptin 2 - Clinformatics; Test type: Other; Hazard Ratio (HR) = 0.85, 95% CI 2-sided [0.65 to 1.10]
Statistical Analysis 3: Comparison: 2nd Gen SUs - Clinformatics vs Linagliptin 3 - Clinformatics; Test type: Other; Hazard Ratio (HR) = 0.65, 95% CI 2-sided [0.49 to 0.86]
Statistical Analysis 4: Comparison: Other DPP-4I - MarketScan vs Linagliptin 1 - MarketScan; Test type: Other; Hazard Ratio (HR) = 0.95, 95% CI 2-sided [0.83 to 1.10]
Statistical Analysis 5: Comparison: Pioglitazone - MarketScan vs Linagliptin 2 - MarketScan; Test type: Other; Hazard Ratio (HR) = 1.01, 95% CI 2-sided [0.85 to 1.19]
Statistical Analysis 6: Comparison: 2nd Gen SUs - MarketScan vs Linagliptin 3 - MarketScan; Test type: Other; Hazard Ratio (HR) = 0.80, 95% CI 2-sided [0.66 to 0.96]

2. Primary Outcome: Number of Participants With Coronary Revascularization
Description: Number of participants with coronary revascularization (elective and non-elective procedure)
Time Frame: Up to 5 years and 7 month
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Other DPP-4I - Clinformatics | Linagliptin 1 - Clinformatics | Pioglitazone - Clinformatics | Linagliptin 2 - Clinformatics | 2nd Gen SUs - Clinformatics | Linagliptin 3 - Clinformatics | Other DPP-4I - MarketScan | Linagliptin 1 - MarketScan | Pioglitazone - MarketScan | Linagliptin 2 - MarketScan | 2nd Gen SUs - MarketScan | Linagliptin 3 - MarketScan
Number analyzed (Participants) | 14688 | 14688 | 10614 | 10614 | 9538 | 9538 | 25135 | 25135 | 18996 | 18996 | 15742 | 15742
Participants | 82 | 81 | 67 | 54 | 67 | 46 | 181 | 181 | 129 | 133 | 125 | 94
Statistical Analysis 1: Comparison: Other DPP-4I - Clinformatics vs Linagliptin 1 - Clinformatics; Test type: Other; Hazard Ratio (HR) = 0.90, 95% CI 2-sided [0.66 to 1.23]
Statistical Analysis 2: Comparison: Pioglitazone - Clinformatics vs Linagliptin 2 - Clinformatics; Test type: Other; Hazard Ratio (HR) = 0.81, 95% CI 2-sided [0.57 to 1.16]
Statistical Analysis 3: Comparison: 2nd Gen SUs - Clinformatics vs Linagliptin 3 - Clinformatics; Test type: Other; Hazard Ratio (HR) = 0.70, 95% CI 2-sided [0.48 to 1.01]
Statistical Analysis 4: Comparison: Other DPP-4I - MarketScan vs Linagliptin 1 - MarketScan; Test type: Other; Hazard Ratio (HR) = 1.04, 95% CI 2-sided [0.85 to 1.28]
Statistical Analysis 5: Comparison: Pioglitazone - MarketScan vs Linagliptin 2 - MarketScan; Test type: Other; Hazard Ratio (HR) = 1.01, 95% CI 2-sided [0.79 to 1.28]
Statistical Analysis 6: Comparison: 2nd Gen SUs - MarketScan vs Linagliptin 3 - MarketScan; Test type: Other; Hazard Ratio (HR) = 0.81, 95% CI 2-sided [0.62 to 1.06]

3. Primary Outcome: Number of Participants With Acute Coronary Syndrome
Description: Number of participants with acute coronary syndrome (ACS). The definition for ACS included acute myocardial infarction (MI), but acute MI was not assessed separately.
Time Frame: Up to 5 years and 7 months
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Other DPP-4I - Clinformatics | Linagliptin 1 - Clinformatics | Pioglitazone - Clinformatics | Linagliptin 2 - Clinformatics | 2nd Gen SUs - Clinformatics | Linagliptin 3 - Clinformatics | Other DPP-4I - MarketScan | Linagliptin 1 - MarketScan | Pioglitazone - MarketScan | Linagliptin 2 - MarketScan | 2nd Gen SUs - MarketScan | Linagliptin 3 - MarketScan
Number analyzed (Participants) | 14688 | 14688 | 10614 | 10614 | 9538 | 9538 | 25135 | 25135 | 18996 | 18996 | 15742 | 15742
Participants | 93 | 72 | 76 | 48 | 72 | 43 | 238 | 221 | 163 | 160 | 161 | 115
Statistical Analysis 1: Comparison: Other DPP-4I - Clinformatics vs Linagliptin 1 - Clinformatics; Test type: Other; Hazard Ratio (HR) = 0.69, 95% CI 2-sided [0.51 to 0.94]
Statistical Analysis 2: Comparison: Pioglitazone - Clinformatics vs Linagliptin 2 - Clinformatics; Test type: Other; Hazard Ratio (HR) = 0.63, 95% CI 2-sided [0.44 to 0.90]
Statistical Analysis 3: Comparison: 2nd Gen SUs - Clinformatics vs Linagliptin 3 - Clinformatics; Test type: Other; Hazard Ratio (HR) = 0.60, 95% CI 2-sided [0.41 to 0.88]
Statistical Analysis 4: Comparison: Other DPP-4I - MarketScan vs Linagliptin 1 - MarketScan; Test type: Other; Hazard Ratio (HR) = 0.97, 95% CI 2-sided [0.81 to 1.17]
Statistical Analysis 5: Comparison: Pioglitazone - MarketScan vs Linagliptin 2 - MarketScan; Test type: Other; Hazard Ratio (HR) = 0.96, 95% CI 2-sided [0.77 to 1.19]
Statistical Analysis 6: Comparison: 2nd Gen SUs - MarketScan vs Linagliptin 3 - MarketScan; Test type: Other; Hazard Ratio (HR) = 0.76, 95% CI 2-sided [0.60 to 0.97]

4. Primary Outcome: Number of Participants With Stroke
Description: Number of participants with ischemic or hemorrhagic stroke. Both types of stroke were included in the definition for stroke, but were not assessed separately
Time Frame: Up to 5 years and 7 months
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Other DPP-4I - Clinformatics | Linagliptin 1 - Clinformatics | Pioglitazone - Clinformatics | Linagliptin 2 - Clinformatics | 2nd Gen SUs - Clinformatics | Linagliptin 3 - Clinformatics | Other DPP-4I - MarketScan | Linagliptin 1 - MarketScan | Pioglitazone - MarketScan | Linagliptin 2 - MarketScan | 2nd Gen SUs - MarketScan | Linagliptin 3 - MarketScan
Number analyzed (Participants) | 14688 | 14688 | 10614 | 10614 | 9538 | 9538 | 25135 | 25135 | 18996 | 18996 | 15742 | 15742
Participants | 42 | 42 | 30 | 30 | 37 | 16 | 113 | 104 | 66 | 74 | 76 | 53
Statistical Analysis 1: Comparison: Other DPP-4I - Clinformatics vs Linagliptin 1 - Clinformatics; Test type: Other; Hazard Ratio (HR) = 0.89, 95% CI 2-sided [0.58 to 1.38]
Statistical Analysis 2: Comparison: Pioglitazone - Clinformatics vs Linagliptin 2 - Clinformatics; Test type: Other; Hazard Ratio (HR) = 0.99, 95% CI 2-sided [0.60 to 1.64]
Statistical Analysis 3: Comparison: 2nd Gen SUs - Clinformatics vs Linagliptin 3 - Clinformatics; Test type: Other; Hazard Ratio (HR) = 0.44, 95% CI 2-sided [0.24 to 0.78]
Statistical Analysis 4: Comparison: Other DPP-4I - MarketScan vs Linagliptin 1 - MarketScan; Test type: Other; Hazard Ratio (HR) = 0.96, 95% CI 2-sided [0.73 to 1.25]
Statistical Analysis 5: Comparison: Pioglitazone - MarketScan vs Linagliptin 2 - MarketScan; Test type: Other; Hazard Ratio (HR) = 1.09, 95% CI 2-sided [0.78 to 1.52]
Statistical Analysis 6: Comparison: 2nd Gen SUs - MarketScan vs Linagliptin 3 - MarketScan; Test type: Other; Hazard Ratio (HR) = 0.74, 95% CI 2-sided [0.52 to 1.05]

5. Secondary Outcome: Number of Participants With Heart Failure Hospitalization
Description: Number of participants with heart failure hospitalization
Time Frame: Up to 5 years and 7 months
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Other DPP-4I - Clinformatics | Linagliptin 1 - Clinformatics | Pioglitazone - Clinformatics | Linagliptin 2 - Clinformatics | 2nd Gen SUs - Clinformatics | Linagliptin 3 - Clinformatics | Other DPP-4I - MarketScan | Linagliptin 1 - MarketScan | Pioglitazone - MarketScan | Linagliptin 2 - MarketScan | 2nd Gen SUs - MarketScan | Linagliptin 3 - MarketScan
Number analyzed (Participants) | 14688 | 14688 | 10614 | 10614 | 9538 | 9538 | 25135 | 25135 | 18996 | 18996 | 15742 | 15742
Participants | 53 | 90 | 27 | 51 | 43 | 47 | 117 | 111 | 58 | 65 | 66 | 49
Statistical Analysis 1: Comparison: Other DPP-4I - Clinformatics vs Linagliptin 1 - Clinformatics; Test type: Other; Hazard Ratio (HR) = 1.55, 95% CI 2-sided [1.10 to 2.18]
Statistical Analysis 2: Comparison: Pioglitazone - Clinformatics vs Linagliptin 2 - Clinformatics; Test type: Other; Hazard Ratio (HR) = 1.90, 95% CI 2-sided [1.19 to 3.03]
Statistical Analysis 3: Comparison: 2nd Gen SUs - Clinformatics vs Linagliptin 3 - Clinformatics; Test type: Other; Hazard Ratio (HR) = 1.11, 95% CI 2-sided [0.73 to 1.68]
Statistical Analysis 4: Comparison: Other DPP-4I - MarketScan vs Linagliptin 1 - MarketScan; Test type: Other; Hazard Ratio (HR) = 0.99, 95% CI 2-sided [0.76 to 1.29]
Statistical Analysis 5: Comparison: Pioglitazone - MarketScan vs Linagliptin 2 - MarketScan; Test type: Other; Hazard Ratio (HR) = 1.10, 95% CI 2-sided [0.77 to 1.56]
Statistical Analysis 6: Comparison: 2nd Gen SUs - MarketScan vs Linagliptin 3 - MarketScan; Test type: Other; Hazard Ratio (HR) = 0.79, 95% CI 2-sided [0.54 to 1.14]

6. Secondary Outcome: Number of Participants With Incident End Stage Renal Disease
Description: Number of participants with incident end stage renal disease (ESRD)
Time Frame: Up to 5 years and 7 months
Population: 1:1 propensity score matched cohorts of linagliptin initiators and comparator groups initiators, identified from Clinformatics and MarketScan database between May 2011 and December 2016. For this outcome only, patients with ESRD at any time prior to and including the day of treatment initiation were excluded.
Measure: Number; unit: Participants
Arm/Group | Other DPP-4I - Clinformatics | Linagliptin 1 - Clinformatics | Pioglitazone - Clinformatics | Linagliptin 2 - Clinformatics | 2nd Gen SUs - Clinformatics | Linagliptin 3 - Clinformatics | Other DPP-4I - MarketScan | Linagliptin 1 - MarketScan | Pioglitazone - MarketScan | Linagliptin 2 - MarketScan | 2nd Gen SUs - MarketScan | Linagliptin 3 - MarketScan
Number analyzed (Participants) | 14472 | 14472 | 10467 | 10467 | 9422 | 9422 | 24714 | 24741 | 18689 | 18689 | 15500 | 15500
Participants | 49 | 75 | 28 | 48 | 38 | 43 | 90 | 116 | 39 | 61 | 53 | 57
Statistical Analysis 1: Comparison: Other DPP-4I - Clinformatics vs Linagliptin 1 - Clinformatics; Test type: Other; Hazard Ratio (HR) = 1.40, 95% CI 2-sided [0.97 to 2.00]
Statistical Analysis 2: Comparison: Pioglitazone - Clinformatics vs Linagliptin 2 - Clinformatics; Test type: Other; Hazard Ratio (HR) = 1.71, 95% CI 2-sided [1.07 to 2.72]
Statistical Analysis 3: Comparison: 2nd Gen SUs - Clinformatics vs Linagliptin 3 - Clinformatics; Test type: Other; Hazard Ratio (HR) = 1.16, 95% CI 2-sided [0.75 to 1.79]
Statistical Analysis 4: Comparison: Other DPP-4I - MarketScan vs Linagliptin 1 - MarketScan; Test type: Other; Hazard Ratio (HR) = 1.34, 95% CI 2-sided [1.01 to 1.76]
Statistical Analysis 5: Comparison: Pioglitazone - MarketScan vs Linagliptin 2 - MarketScan; Test type: Other; Hazard Ratio (HR) = 1.52, 95% CI 2-sided [1.02 to 2.27]
Statistical Analysis 6: Comparison: 2nd Gen SUs - MarketScan vs Linagliptin 3 - MarketScan; Test type: Other; Hazard Ratio (HR) = 1.17, 95% CI 2-sided [0.81 to 1.71]

7. Secondary Outcome: Number of Participants With Acute Renal Failure
Description: Number of participants with acute renal failure
Time Frame: Up to 5 years and 7 months
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Other DPP-4I - Clinformatics | Linagliptin 1 - Clinformatics | Pioglitazone - Clinformatics | Linagliptin 2 - Clinformatics | 2nd Gen SUs - Clinformatics | Linagliptin 3 - Clinformatics | Other DPP-4I - MarketScan | Linagliptin 1 - MarketScan | Pioglitazone - MarketScan | Linagliptin 2 - MarketScan | 2nd Gen SUs - MarketScan | Linagliptin 3 - MarketScan
Number analyzed (Participants) | 14688 | 14688 | 10614 | 10614 | 9538 | 9538 | 25135 | 25135 | 18996 | 18996 | 15742 | 15742
Participants | 222 | 300 | 152 | 198 | 163 | 167 | 433 | 430 | 240 | 263 | 238 | 200
Statistical Analysis 1: Comparison: Other DPP-4I - Clinformatics vs Linagliptin 1 - Clinformatics; Test type: Other; Hazard Ratio (HR) = 1.24, 95% CI 2-sided [1.04 to 1.47]
Statistical Analysis 2: Comparison: Pioglitazone - Clinformatics vs Linagliptin 2 - Clinformatics; Test type: Other; Hazard Ratio (HR) = 1.31, 95% CI 2-sided [1.06 to 1.61]
Statistical Analysis 3: Comparison: 2nd Gen SUs - Clinformatics vs Linagliptin 3 - Clinformatics; Test type: Other; Hazard Ratio (HR) = 1.04, 95% CI 2-sided [0.84 to 1.29]
Statistical Analysis 4: Comparison: Other DPP-4I - MarketScan vs Linagliptin 1 - MarketScan; Test type: Other; Hazard Ratio (HR) = 1.04, 95% CI 2-sided [0.91 to 1.19]
Statistical Analysis 5: Comparison: Pioglitazone - MarketScan vs Linagliptin 2 - MarketScan; Test type: Other; Hazard Ratio (HR) = 1.07, 95% CI 2-sided [0.90 to 1.27]
Statistical Analysis 6: Comparison: 2nd Gen SUs - MarketScan vs Linagliptin 3 - MarketScan; Test type: Other; Hazard Ratio (HR) = 0.91, 95% CI 2-sided [0.75 to 1.09]

8. Secondary Outcome: Number of Participants With Acute Renal Failure Requiring Dialysis
Description: Number of patients with acute renal failure requiring dialysis
Time Frame: Up to 5 years and 7 months
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Other DPP-4I - Clinformatics | Linagliptin 1 - Clinformatics | Pioglitazone - Clinformatics | Linagliptin 2 - Clinformatics | 2nd Gen SUs - Clinformatics | Linagliptin 3 - Clinformatics | Other DPP-4I - MarketScan | Linagliptin 1 - MarketScan | Pioglitazone - MarketScan | Linagliptin 2 - MarketScan | 2nd Gen SUs - MarketScan | Linagliptin 3 - MarketScan
Number analyzed (Participants) | 14688 | 14688 | 10614 | 10614 | 9538 | 9538 | 25135 | 25135 | 18996 | 18996 | 15742 | 15742
Participants | 7 | 13 | 6 | 10 | 5 | 9 | 14 | 16 | 9 | 9 | 7 | 11
Statistical Analysis 1: Comparison: Other DPP-4I - Clinformatics vs Linagliptin 1 - Clinformatics; Test type: Other; Hazard Ratio (HR) = 1.62, 95% CI 2-sided [0.64 to 4.06]
Statistical Analysis 2: Comparison: Pioglitazone - Clinformatics vs Linagliptin 2 - Clinformatics; Test type: Other; Hazard Ratio (HR) = 1.67, 95% CI 2-sided [0.61 to 4.58]
Statistical Analysis 3: Comparison: 2nd Gen SUs - Clinformatics vs Linagliptin 3 - Clinformatics; Test type: Other; Hazard Ratio (HR) = 1.84, 95% CI 2-sided [0.62 to 5.48]
Statistical Analysis 4: Comparison: Other DPP-4I - MarketScan vs Linagliptin 1 - MarketScan; Test type: Other; Hazard Ratio (HR) = 1.17, 95% CI 2-sided [0.57 to 2.40]
Statistical Analysis 5: Comparison: Pioglitazone - MarketScan vs Linagliptin 2 - MarketScan; Test type: Other; Hazard Ratio (HR) = 0.96, 95% CI 2-sided [0.38 to 2.43]
Statistical Analysis 6: Comparison: 2nd Gen SUs - MarketScan vs Linagliptin 3 - MarketScan; Test type: Other; Hazard Ratio (HR) = 1.65, 95% CI 2-sided [0.64 to 4.27]

ADVERSE EVENTS:
Description: As this is a non-interventional study with secondary use of data retrieved from a US health claims database, safety monitoring and safety reporting on an individual case level is not applicable.
Arm/Group | Other DPP-4I - Clinformatics | Linagliptin 1 - Clinformatics | Pioglitazone - Clinformatics | Linagliptin 2 - Clinformatics | 2nd Gen SUs - Clinformatics | Linagliptin 3 - Clinformatics | Other DPP-4I - MarketScan | Linagliptin 1 - MarketScan | Pioglitazone - MarketScan | Linagliptin 2 - MarketScan | 2nd Gen SUs - MarketScan | Linagliptin 3 - MarketScan
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
Pioglitazone is contraindicated among patients with heart failure and edema. This suggests pioglitazone may not be a proper comparator in the assessment of the association between linagliptin and heart failure hospitalization or renal outcomes.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2014-07-03): https://cdn.clinicaltrials.gov/large-docs/78/NCT02197078/Prot_SAP_000.pdf